CLINICAL TRIAL: NCT00806221
Title: An Open-Label Study Investigating the Effects of Early Skin Barrier Protection on the Development of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Eric Simpson, Professor, Dermatology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00002726
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Prevention; Skin Barrier
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Emollients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emollient (Experimental): Skin barrier protection from birth
  Interventions: Drug: emollient (Cetaphil cream)

INTERVENTIONS:
Drug: emollient (Cetaphil cream) — Cetaphil cream applied daily from birth

SUMMARY:
The purpose of this study is to determine whether early use of a bland emollient in newborns, prior to the clinical signs of skin disease, will delay the onset or prevent the development of atopic dermatitis.

DETAILED DESCRIPTION:
All neonates will be treated with Cetaphil cream starting within 1 week of birth. All neonates enrolled will have an increased risk of developing atopic dermatitis because they have a family history of either asthma, hay fever, or atopic dermatitis. These neonates will then be followed for 2 years for the signs and symptoms of atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* at least one parent diagnosed with Atopic Dermatitis
* one parent or sibling with hayfever or asthma

Exclusion Criteria:

* newborns with dermatitis at birth
* newborns born greater than four weeks prematurely
* newborns with medical problems necessitating prolonged hospitalization
* newborns diagnosed with any immune deficiency syndrome

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Department of Dermatology, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emollient
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Emollient
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  gender/sex was not recorded | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic Caucasian | 16
  Hispanic Caucasian | 2
  Asian | 2
  African American | 2
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Skin Irritation
Time Frame: 1 and 2 year time points
Measure: Count of Participants; unit: Participants
Arm/Group | Emollient
Number analyzed (Participants) | 22
Participants | 0

2. Primary Outcome: Incidence of Skin Infection
Time Frame: 1 and 2 year timepoints
Measure: Count of Participants; unit: Participants
Arm/Group | Emollient
Number analyzed (Participants) | 22
Participants | 0

3. Primary Outcome: Compliance With Protocol
Time Frame: over two years
Measure: Number; unit: participants
Arm/Group | Emollient
Number analyzed (Participants) | 22
participants | 20

4. Secondary Outcome: Development of Eczema
Time Frame: 1 and 2 year time points
Measure: Count of Participants; unit: Participants
Arm/Group | Emollient
Number analyzed (Participants) | 22
Participants | 5

ADVERSE EVENTS:
Arm/Group | Emollient
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No